CLINICAL TRIAL: NCT06815679
Title: The Physiological Effects of Nebulized Salbutamol in Patients With Acute Respiratory Failure During HFNC
Brief Title: Physiological Effects of Nebulized Salbutamol in Acute Respiratory Failure Patients on HFNC
Acronym: PENSAFE-HFNC
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Aerogen (Industry)
Responsible Party: Principal Investigator, Savino Spadaro, Professor, Università degli Studi di Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nebulized Salbutamol and HFNC
Record Dates: First submitted 2025-01-09; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Acute Respiratory Failure; Pneumonia
Keywords: salbutamol; acute respiratory failure; high flow nasal cannalae; aerosol delivery
MeSH Terms: conditions — Pneumonia | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salbutamol (Experimental): All patients will received ventilatory support with HFNC by adjusting gas flows to 30 L/min with 100% relative humidity, heated to 37 C, adjusting FiO2 levels to maintain SpO2 between 92 and 96%. After 20 min, each patient remaining on ventilatory support with HFNC will receive administration of salbutamol 2.5 mg via the vibrating mesh nebulizer (VMN) (Aerogen Solo®, Aerogen Ltd., Galway, Ireland) positioned immediately downstream of the humidification chamber of the HFNC system, using the dedicated connector.
  Interventions: Drug: salbutamol 2.5 mg via vibrating mesh nebulizer (VMN)

INTERVENTIONS:
Drug: salbutamol 2.5 mg via vibrating mesh nebulizer (VMN) — To evaluate the patient's respiratory effort, the pressure-time product (PTPes) and the delta of Pes oscillations during inspiration (∆ Pes) will be obtained from the analysis of the Pes curve. Global and regional pulmonary tidal volumes will be evaluated with Electrical Impedance Tomography

SUMMARY:
This is a prospective physiological interventional study that assess the feasibility and safety of administering salbutamol using a vibrating mesh nebulizer during HFNC in patients with acute hypoxemic respiratory failure (AHRF). We evaluate whether this method of salbutamol delivery can reduce inspiratory effort and improve global and regional lung ventilation in AHRF patients. To achieve this, the study will record and analyze the following: esophageal pressure (Pes) curves, global and regional tidal volumes, minute ventilation, and changes in global and regional lung ventilation assessed through Electrical Impedance Tomography (EIT).

DETAILED DESCRIPTION:
To evaluate the patient's respiratory effort, the pressure-time product (PTPes) and the delta of Pes oscillations during inspiration (∆ Pes) will be obtained from the analysis of the Pes curve. Global and regional pulmonary tidal volumes will be evaluated with EIT.

ELIGIBILITY:
Inclusion Criteria:

* • Age > 18, < 90 years

  * Non-intubated critically ill patients with AHRF due to pneumonia (diagnosis is based on the presence of infiltrates on chest X-ray and the onset of clinical signs of infection less than 7 days earlier)
  * PaO2/FiO2 ≤ 300 mmHg
  * Patients receiving oxygen therapy

Exclusion Criteria:

* • Age < 18 years

  * Hypercapnia (PaCO2 > 50 mmHg)
  * Hemodynamic instability (Systolic blood pressure < 90 mmHg or Mean arterial pressure < 60 or high dose of vasoactive drugs)
  * Tachycardia or tachyarrhythmia (HR > 130 b/min)
  * Known allergy or intolerance to salbutamol
  * Patient has received inhaled therapy with short-acting beta 2 agonists < 8 hours before or with long-acting beta 2 agonists < 24 hours before
  * Acute exacerbation of COPD or bronchial asthma
  * Cardiogenic pulmonary edema
  * GCS ≤ 12
  * Contraindication for EIT (e.g. ICD)
  * Pregnancy
  * Patient refuses to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the changes of inspiratory effort based on the analysis of the oesophageal pressure curve. | The measurement of ΔPes will be conducted: After 20 minutes of ventilatory support with HFNC (Time 0) 10 minutes following the completion of Salbutamol administration (Time 1) At 1 hour, 2 hours, and 3 hours post-Salbutamol administration
  Our hypothesis is based on changes of inspiratory effort, based on the analysis of the delta esophageal pressure (ΔPes), after the administration of Salbutamol by via a vibrating mesh nebulizer during HFNC in patients with AHRF. Evaluating the delta esophageal pressure (ΔPes) requires careful measurement of esophageal pressure (Pes) during the respiratory cycle. ΔPes specifically reflects the inspiratory effort or the work of breathing (WOB), as it measures the difference between the maximum inspiratory and expiratory Pes values during each breath.

SECONDARY OUTCOMES:
Feasibility and safety of administering salbutamol via a vibrating mesh nebulize | Data Collection Points: Baseline (prior to Salbutamol administration). During nebulization. Post-nebulization at 10 minutes, 1 hour, 2 hours, and 3 hours.
  To evaluate the feasibility and safety of administering salbutamol via a vibrating mesh nebulizer during HFNC in patients with AHRF. The safety evaluation involves identifying and mitigating potential risks associated with the intervention.
  Monitor patients for known side effects of Salbutamol, such as:
  Tachycardia (>100bpm) Arrhythmias (identified by bpm; millisecond)
  Continuously monitor:
  Heart rate (to detect tachycardia; bpm)
Feasibility and safety of administering salbutamol via a vibrating mesh nebulize To evaluate the feasibility and safety of administering salbutamol via a vibrating mesh nebulizer during HFNC in patients with AHRF. The safety evaluation involves identif | Data Collection Points: Baseline (prior to Salbutamol administration). During nebulization. Post-nebulization at 10 minutes, 1 hour, 2 hours, and 3 hours.
  To evaluate the feasibility and safety of administering salbutamol via a vibrating mesh nebulizer during HFNC in patients with AHRF. The safety evaluation involves identifying and mitigating potential risks associated with the intervention. Hypokalemia (definied <3.0 to 3.4 mEq/L)
Feasibility and safety of administering salbutamol via a vibrating mesh nebulize | [Time Frame: Data Collection Points: Baseline (prior to Salbutamol administration). During nebulization. Post-nebulization at 10 minutes, 1 hour, 2 hours, and 3 hours.]
  To evaluate the feasibility and safety of administering salbutamol via a vibrating mesh nebulizer during HFNC in patients with AHRF. The safety evaluation involves identifying and mitigating potential risks associated with the intervention. Record any exacerbation of respiratory distress or intolerance to the nebulization process. Continuously monitor: Oxygen saturation (SpO₂,%) and respiratory rate (to ensure adequate oxygenation and ventilation)
Feasibility and safety of administering salbutamol via a vibrating mesh nebulize | : Baseline (prior to Salbutamol administration). During nebulization. Post-nebulization at 10 minutes, 1 hour, 2 hours, and 3 hours.]
  To evaluate the feasibility and safety of administering salbutamol via a vibrating mesh nebulizer during HFNC in patients with AHRF. Patient Tolerance: Document patient comfort scale (from 1 to 10)
Evaluation of global and regional ventilation by EIT | Data Collection Points: Baseline (before Salbutamol administration) during HFNC therapy. Post-Salbutamol: 10 minutes (early phase of response) 1 hour, 2 hours, and 3 hours after Salbutamol administration.
  To evaluate the improvement of global and regional ventilation based on data obtained with EIT after the administration of salbutamol via a vibrating mesh nebulizer during HFNC in patients with AHRF. EIT provides real-time, non-invasive monitoring of ventilation by measuring regional changes in electrical impedance within the thorax. Parameters to Monitor with EIT: Global Ventilation: Overall changes in lung ventilation during tidal breathing.
  Regional Ventilation Distribution in percentage in tidal volume (%).
Evaluation of global and regional ventilation by EIT | Data Collection Points: Baseline (before Salbutamol administration) during HFNC therapy. Post-Salbutamol: 10 minutes (early phase of response) 1 hour, 2 hours, and 3 hours after Salbutamol administration.
  To evaluate the improvement of regional ventilation based on data obtained with EIT after the administration of salbutamol via a vibrating mesh nebulizer during HFNC in patients with AHRF. Regional Ventilation Delay (RVD) Definition: Measures the time delay in the filling of different lung regions during inhalation.
  Unit: Milliseconds (ms) or as a percentage of the respiratory cycle.
Evaluation of global and regional ventilation by EIT | Data Collection Points: Baseline (before Salbutamol administration) during HFNC therapy. Post-Salbutamol: 10 minutes (early phase of response) 1 hour, 2 hours, and 3 hours after Salbutamol administration.
  To evaluate the improvement of regional ventilation based on data obtained with EIT after the administration of salbutamol via a vibrating mesh nebulizer during HFNC in patients with AHRF. Center of Ventilation (CoV) Definition: Describes the gravity-dependent distribution of ventilation from ventral (front) to dorsal (back) lung regions.
  Unit: Percentage (%), representing the shift in ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Alberto Volta, Professor, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Azienda ospedaliera Universitaria di Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] MacLoughlin R, Mac Giolla Eain M. Performance Characterisation of the Airvo2TM Nebuliser Adapter in Combination with the Aerogen SoloTM Vibrating Mesh Nebuliser for in Line Aerosol Therapy during High Flow Nasal Oxygen Therapy. Pharmaceutics. 2024 Apr 20;16(4):565. doi: 10.3390/pharmaceutics16040565. PMID 38675226
- [Result] Calabrese C, Annunziata A, Mariniello DF, Allocca V, Imitazione P, Cauteruccio R, Simioli F, Fiorentino G. Aerosol delivery through high-flow nasal therapy: Technical issues and clinical benefits. Front Med (Lausanne). 2023 Jan 18;9:1098427. doi: 10.3389/fmed.2022.1098427. eCollection 2022. PMID 36743674
- [Result] Arunsurat I, Rittayamai N, Chuaychoo B, Tangchityongsiva S, Promsarn S, Yuenyong S, Chow CW, Brochard L. Bronchodilator Efficacy of High-Flow Nasal Cannula in COPD: Vibrating Mesh Nebulizer Versus Jet Nebulizer. Respir Care. 2024 Jan 24;69(2):157-165. doi: 10.4187/respcare.11139. PMID 37607815